CLINICAL TRIAL: NCT04802902
Title: Feasibility of Immunotherapy Plus Chemotherapy Administration to Patients With Bronchial Cancer in a Hospital-at- Home Setting - CombHADom
Brief Title: Feasibility of Immunotherapy Plus Chemotherapy Administration to Patients With Bronchial Cancer in a Hospital-at- Home Setting
Acronym: CombHADom
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Other Study IDs: CHPAU2021/03
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Bronchial Cancer
Keywords: immunotherapy; chimiotherapy; Bronchial cancer; home-based hospitalization
MeSH Terms: conditions — Carcinoma, Bronchogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: home-based hospitalization — management in a hospital-at-home programme of patients treated by immunotherapy and chimiotherapy combo for bronchial cancer

SUMMARY:
This observational prospective monosite study aims to describe, for the first time, management in a hospital-at-home programme of patients treated by immunotherapy-chemotherapy combo for bronchial cancer in maintenance phase of first row metastatic treatment.

The feasibility in good conditions of this management, the patients' quality of life and their satisfaction will be evaluated. A cost-benefit analysis will be done to compare hospital-at-home programme and classical day hospitalization.

DETAILED DESCRIPTION:
Those last years, immunotherapy treatment for bronchial cancers allowed considerable progress in terms of tumoral answer, survival without progression and global survival. Usually administered in the day hospitalization department, its preparation and administration to the patient are compatible with hospital-at-home management. This type of management has particularly developed in the context of the COVID pandemic and recommendations for good practices in hospital-at-home immunotherapy have recently been drafted by FITC (Société Française d'Immuno-Thérapie du Cancer). These recommendations open the way for administration of immunotherapy and chemotherapy combo in hospital-at-home. At the moment, there is no study stating the feasibility of home hospitalization for patients treated by immunotherapy-chemotherapy combo. To follow up on the feasibility study of home immunotherapy (ImHADom) carried out at CH Pau from March 2019 to March 2021, the sponsor propose to evaluate with descriptive study the feasibility under the same conditions of chemotherapy-immunotherapy in patients treated in the maintenance phase of a first metastatic row.

This study will be proposed to all the patients in maintenance phase of first row treatment with at least one positive tumoral imaging assessment (stable disease or partial response) for whom home hospitalization has been decided and scheduled by the healthcare team in a medical staff meeting.

The patients included in the study will be followed according to the common practice: a consultation every 3 months during 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over,
* with bronchial metastatic cancer treated in first row maintenance phase by immunotherapy-chemotherapy combo,
* having at least one assessments of the response to immunotherapy received in day hospitalization with efficiency (stability or partial response),
* without any graded higher than 1 adverse effects, or uncontrolled grade 1 adverse effects related to immunotherapy
* eligible for a home-based hospitalization

Exclusion Criteria:

* Frail patients requiring a frequent medical assessment thus day hospitalization cares

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by immunotherapy and chemotherapy combo in maintenance phase for bronchial cancer
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of home-based immunotherapy (percentage of patients who interrupted their home hospitalization for reasons directly linked to that management) | 1 year
  Feasibility under good conditions of home-based immunotherapy, defined by the percentage of patients who interrupted their home hospitalization for reasons directly linked to that management.

SECONDARY OUTCOMES:
Cost-benefit analysis | 1 year
  A cost-benefit analysis comparing hospital-at-home programme and classical day hospitalization
Number of adverse effects occuring during the study | 1 year
  Immunotherapy related adverse effects monitoring criteria evaluation
Number of Incidents occurring during the Hospital at Home program handling process | 1 year
  The occurrence of possible incidents related to the Hospital at Home program will be collected at each home based hospitalization.
Quality of Life Questionnaire (EORTC QLQ-C30) total score | at inclusion, month 3, 6 9 and 12
  To study the patient's reported quality of life before and throughout therapy. Quality of life score obtained through self-administered EORCT QLQ-C30 questionnaire at inclusion, month 3, 6 9 and 12.
Patients' Satisfaction Questionnaire | at month 3, 6 9 and 12
  Patients' satisfaction with their home base management will be assessed with a questionnaire. It will be collected at month 3, 6 9 and 12
Healthcare professional satisfaction | at month 6, 12, 18 and 24 of the study
  Healthcare professional satisfaction will be assessed with a questionnaire. It will be collected at month 6, 12, 18 and 24 of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier de pau, Pau, Aquitaine, France